CLINICAL TRIAL: NCT01484795
Title: Non Invasive Ventilation in Acute Myocardial Infarction
Brief Title: Noninvasive Ventilation in Acute Myocardial Infarction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Cristina Marcia Dias, PhD, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Cristina Dias
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Acute Myocardial Infarction
Keywords: noninvasive ventilation; autonomic nervous system

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous positive airway pressure (Experimental)
  Interventions: Device: Continuos positive airway pressure (Respironics)
- BILEVEL (Experimental)
  Interventions: Device: BILEVEL (Respironics)

INTERVENTIONS:
Device: BILEVEL (Respironics) — Bilevel was delivered by a Bipap® ventilator (Respironics Inc, Murrysville, PA), applied via facial mask, with inspiratory positive pressure (IPAP) of 20 cmH2O and expiratory positive airway pressure (EPAP) of 10 cmH2O.
  Other Names: BIPAP
  Arms: BILEVEL
Device: Continuos positive airway pressure (Respironics) — CPAP was delivered by a ventilator (Respironics Inc, Murrysville, PA), applied via a facial mask, with expiratory positive airway pressure of 10 cmH2O.
  Other Names: CPAP
  Arms: Continuous positive airway pressure

SUMMARY:
Cardiovascular diseases, especially acute myocardial infarction (AMI), represent the major cause of mortality and morbidity in the world. The myocardial ischemia is often the precipitating cause of pulmonary edema and noninvasive ventilation (NIV) with positive pressure has been used as a therapeutic modality.

Objective: to evaluate the effects of NIV on heart rate variability (HRV) and on ventilatory and hemodynamic variables in patients with myocardial infarction.

Materials and methods: ten patients with acute myocardial infarction, with Killip I classification, will use continuous positive airway pressure (CPAP) and Bilevel ventilation during 30 minutes, according randomization. Then ventilatory and hemodynamic variables will be registered and electrocardiogram signals will be recorded for posterior analyses of HRV. Data will be collected before, during and after positive pressure ventilation.

Statistical Analysis: Data will be compared using One Way Anova Repeated Measures, followed by Tukey test.

DETAILED DESCRIPTION:
The patients will be recruited in Bonsucesso Federal Hospital with diagnosis of myocardial infarction, confirmed by electrocardiogram and cardiac enzymes, between 24 and 72 hours after the event.

Participation in the study protocol will be done according to eligibility criteria:

The study will be a randomized and crossover clinical trial for evaluation and comparison of heart rate variability and ventilatory and hemodynamics variables during ventilation with CPAP and Bilevel.

CPAP will be applied via a facial mask, with expiratory positive airway pressure of 10 cmH2O. Bilevel will be applied via facial mask, with inspiratory positive pressure (IPAP) of 20 cmH2O and expiratory positive airway pressure (EPAP) of 10 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction with Killip I classification, hemodynamic stability, between 24 and 72 hours post event;
* agreement to participate in the study, according written informed consent;
* 45 to 80 years old age.

Exclusion Criteria:

* unstable angina;
* systolic blood pressure < 80 mmHg;
* patients who presented ST elevation > 2 mm or with second-degree atrioventricular block;
* presence of pacemaker.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
evaluate HRV during NIV after acute myocardial infarction | six months
  The study consisted of randomized and crossover clinical trial for evaluation and comparison of heart rate variability and ventilatory and hemodynamics variables during ventilation with CPAP and Bilevel.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Dias, PT - PhD, Principal Investigator — Centro Universitário Augusto Motta